CLINICAL TRIAL: NCT04064021
Title: Clinical Trial to Measure Efficacy of Acupuncture Treatment for Alzheimer's Dementia as Measured by MOCA(Montreal Cognitive Assessment)
Brief Title: Acupuncture Treatment for Improving Alzheimer's Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to covid19 pandemic
Sponsor: N & S Neurology Center, A Medical Group, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS1
Record Dates: First submitted 2015-04-28; First posted 2019-08-21 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Cognitive Deficits; Alzheimer Disease
Keywords: Acupunture
MeSH Terms: conditions — Cognition Disorders; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture (Experimental): Acupuncture 12 sessions over 6 week to be given to pateints
  Interventions: Procedure: Acupunture

INTERVENTIONS:
Procedure: Acupunture — Patient will receive 12 acupuncture treatments over 6 weeks (2x per week)

SUMMARY:
Evaluate cognitive improvement pre amd post acupuncture treatment in patients with probable alzheimer's dementia as measured by MOCA score and also per form A( measure of patient's personal information). Also caregiver input.

DETAILED DESCRIPTION:
Patient's with diagnosis of probable mild to moderate AD will be enrolled in this study. Patient will undergo neurological examination including MOCA. Examiner will also fill out Form A at the time of initial evaluation.

Patient will then undergo series of acupuncture treatments 2 per week for 6 weeks(12 acupuncture treatment). At end of this intervention patients will be reassessed using same testing(MOCA and form A) Data collected will be assessed via statistical analysis to see if there is any statistically significant improvement.

Acupuncture points used in this trial will stay the same for all subjects and throughout the course. The points will be Si Shen Chong, ST36, 37, LV 2,3,6, GB 34, 39, Xia San Huang, LI 11, LI 4.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate AD

Exclusion Criteria:

* Severe AD

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Improvement on Montreal Cognitive Assessment test of 5 points or more than baseline( total score is out of 30 points) | 12 weeks
  Subject will complete 3 MOCA assessment prior to study over 1 week time. Best score of three is used.
  After study is complete subject will also undergo 3 MOCA assessment over 1 week immediately after study. Again best score is used.

SECONDARY OUTCOMES:
Improvement of Montreal Cognitive Assessment test by category than raw total score | 12 weeks
  performance on various subcategory will also be reviewed to see if one category improves over other category. (Example: Visual-spacial parameters improves over language)

CONTACTS AND LOCATIONS:
Overall Officials: SANJAY CHAUHAN, M.D., Principal Investigator — N & S Neurology Center, A Medical Group, Inc